CLINICAL TRIAL: NCT02963688
Title: Prevalence Study of Germline and/or Somatic BRCA1/2 Mutation in Korean Patients With High-Grade Serous and/or Endometrioid Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: BRCA 1/2 Mutation in Korean Patients With Epithelial Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: SMC 2015-05-064
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: To Investigate the Prevalence of BRCA 1/2 Mutation Among Ovarian Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- KGOG 3019: Korean women with HG serous and/or endometrioid epithelial ovarian cancer
  Interventions: Genetic: Ion AmpliSeq BRCA 1/2 Panel (Life Technologies, Carlsbad, CA, USA) ,Ion PGM platform

INTERVENTIONS:
Genetic: Ion AmpliSeq BRCA 1/2 Panel (Life Technologies, Carlsbad, CA, USA) ,Ion PGM platform — BRCA1,2 Germline /Somatic mutation test

SUMMARY:
PURPOSE: To investigate the prevalence and clinical correlation of the germline BRCA 1/2 mutation in Korean patients with high grade(HG) serous and/or endometrioid epithelial ovarian cancer (EOC).

PATIENTS AND METHODS: In a nationwide case-control study on EOC conducted in Korea between 2010 and 2015, 298 Korean women with HG serous and/or endometrioid EOC were tested for gBRCA 1/2 mutation, regardless of the family history. Mutation screening was performed using the Ion AmpliSeq BRCA 1/2 Panel (Life Technologies, Carlsbad, CA, USA) and Ion PGM platform according to the manufacturer's instructions. Clinical characteristics including survival outcome was assessed in gBRCAm carriers.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years of age and older with previously untreated, HG serous and/or endometrioid EOC, fallopian tube or primary peritoneal carcinoma who consented to genetic testing between 2010 and 2015

Exclusion Criteria:

* women with mucinous , clear cell, low-grade serous or endometrioid, mixed epithelial adenocarcinoma, undiffereniated carcinoma or malignant brenner's tumor

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women 18 years of age and older with previously untreated, HG serous and/or endometrioid EOC, fallopian tube or primary peritoneal carcinoma who consented to genetic testing between 2010 and 2015
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of positive mutation among ovarian cancer patients | 5 year

IPD SHARING:
Plan to Share IPD: No